## STATISTICAL ANALYSIS PLAN

Fitforlife; Peer-mentor driven physical exercise for persons affected by psychosis.

1.6.2019

## Statistical analysis plan

Baseline descriptions will be presented and used in the different analyses to see if gender, duration of psychosis, neuroleptics affects the different outcomes.

The main outcome social function will be analyzed using  $\chi^2$  tests and analysis of variance for categorical outcomes using data from baseline to 6 months. Pre- to post-intervention (withingroup) analyses will be performed using paired-sample *t*tests, with effect sizes (Hedges' *g*) calculated for statistically significant values. The participants will be divided according to attended number of training sessions. This will be done in quartiles and used to look at between group differences (analysis of covariance- ANCOVA). A sub analysis will be done including those with accelerometer data from the entire study period. Baseline score will be included as covariates in each model.

Parametric test assumptions will be checked before running all analyses. Normality will be assessed using the Shapiro–Wilks test and normal probability plot, and homogeneity of variance using Levene's test. For analyses involving unequal sample sizes, Welch's test might be considered. Similar procedures will be used when analyzing blood samples, inflammatory and metabolic markers as well as cognitive test data. Normative data from the cog state data base will be used for comparison. Multilevel analysis will be used taking into account the included open care units.